CLINICAL TRIAL: NCT02270047
Title: SATIN The Acute Effect of Orange Nectar With NAXUS Fibre Made by Novel Processing on Satiety and Satiation
Acronym: SATIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Leeds (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Anders Mikael Sjödin, MD, PHD ass professor, Associated Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B315
Record Dates: First submitted 2014-10-13; First posted 2014-10-21 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Appetite
Keywords: Ad libitum energy intake; Appetite sensation
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Orange nectar with NAXUS fibre, 5g/100mL
  Interventions: Dietary Supplement: Orange Nectar with fibre
- B (Placebo Comparator): Orange nectar
  Interventions: Dietary Supplement: Orange nectar

INTERVENTIONS:
Dietary Supplement: Orange nectar — Orange nectar
  Arms: B
Dietary Supplement: Orange Nectar with fibre
  Arms: A

SUMMARY:
A 4 week double blinded parallel design with an intervention condition and a control condition will be employed. After having completed screening procedure and a baseline test day, participants will be randomized to either intervention or control condition. In the following 4 weeks, the participants will have to consume the distributed food product daily before completing another test day.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* BMI between 23.0-27.9 kg/m2
* Regular breakfast eaters (eating breakfast ≥ 4 times a week)
* Regular menstrual periods

Exclusion Criteria:

* Significant health problems as judged by the investigator
* Taking any medication or supplements known to affect appetite or body weight within the past month and/or during the study as judged by the investigator
* Pregnant, planning to become pregnant within the next 4 weeks or breastfeeding
* History of anaphylaxis to food
* Any known food allergies or food intolerance, specifically the below listed:

  1. Cereals containing gluten, namely: wheat, rye, barley, oats, spelt, kamut or their hybridised strains, and products thereof;
  2. Crustaceans and products thereof;
  3. Eggs and products thereof;
  4. Fish and products thereof;
  5. Peanuts and products thereof;
  6. Soybeans and products thereof;
  7. Milk and products thereof (including lactose);
  8. Nuts, namely: almonds (Amygdalus communis L.), hazelnuts (Corylus avellana), walnuts (Juglans regia), cashews (Anacardium occidentale), pecan nuts (Carya illinoinensis (Wangenh.) K. Koch), Brazil nuts (Bertholletia excelsa), pistachio nuts (Pistacia vera), macadamia or Queensland nuts (Macadamia ternifolia), and products thereof, except for nuts used for making alcoholic distillates including ethyl alcohol of agricultural origin;
  9. Celery and products thereof;
  10. Mustard and products thereof;
  11. Sesame seeds and products thereof;
  12. Sulphur dioxide and sulphites;
  13. Lupin
  14. Molluscs
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes)
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Significant changes in physical activity patterns in the past 4 weeks or intention to change during the study as judged by the investigator
* Significant change in diet in the past 4 weeks or intention to change the diet during the study as judged by the investigator
* Use of systemic or local treatment likely to interfere with evaluation of the study parameters as judged by the investigator
* Participants who work in appetite or feeding related areas
* Participants not able to comply with the study protocol
* Post-menopausal

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
AD libitum energy intake | week0, week 4

SECONDARY OUTCOMES:
VAS score for appetite sensation | Week 0, week 4
  Perceptions of hunger, fullness, desire to eat, prospective consumption will be assessed using 100 mm VAS scales

OTHER OUTCOMES:
Eating behaviour | week 0 week 4
  Eating behaviour will be assessed by the binge eating scale from Gormally et al. 1982, the Control og Eating questionnaire by Hill et al. 1991, the Power og food scale by Lowe et al 2009, and the Three Factor Eating Questionnaire by Stunkard and Messick, 1985

CONTACTS AND LOCATIONS:
Overall Officials: Graham Finlayson, Ass Prof, Principal Investigator — University of Liverpool
Locations (1):
- Department of Nutrition Exercise and Sports, Copenhagen, Copenhagen, Denmark